CLINICAL TRIAL: NCT05293132
Title: The Effect of Montelukast Versus Co Enzyme Q10 on the Clinical Outcome of Patients With Sepsis
Brief Title: Effect of Montelukast Versus Co Enzyme in Sepsis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada Hussein, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC # 50
Record Dates: First submitted 2022-02-18; First posted 2022-03-24 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — montelukast; coenzyme Q10

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Montelukast group (Experimental): 30 patients will receive montelukast sodium 10 mg/day film coated tablets (Singulair®; Merck & Co Inc) or (Clear air®; Amoun Pharmaceutical Company S.A.E., Egypt) in addition to the standard sepsis treatment starting from the onset of the diagnosis of sepsis till discharge from ICU, or death.
  Interventions: Drug: Montelukast Sodium 10 mg; Drug: Standard Treatment
- Co Enzyme Q10 group (Experimental): 30 patients will receive co enzyme Q10 capsule 210 mg / day (MEPACO Pharmaceutical Company (Egypt) in addition to the standard sepsis treatment starting from the onset of the diagnosis of sepsis till discharge from ICU, or death.
  Interventions: Drug: Co-Enzyme Q10; Drug: Standard Treatment
- Control group (Active Comparator): 30 patients will receive the standard treatment of sepsis from the onset of the diagnosis of sepsis till discharge from ICU, or death.
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Drug: Montelukast Sodium 10 mg — Film coated tablets containing 10 mg montelukast
  Other Names: (Singulair®; Merck & Co Inc) or (Clear air®; Amoun Pharmaceutical Company S.A.E., Egypt)
  Arms: Montelukast group
Drug: Co-Enzyme Q10 — Capsules contain 210 mg Co-Enzyme Q10
  Other Names: Co enzyme Q10(MEPACO Pharmaceutical Company (Egypt)
  Arms: Co Enzyme Q10 group
Drug: Standard Treatment — Standard sepsis treatment includes fluid resuscitation, early administration of intravenous broad spectrum antibiotic (ceftriaxone 2gm/24 hour or meropenem 1g/8 hours, linezolid 600/12hours) till obtaining the microbiological culture to narrow the coverage, paracetamol intravenous antipyretic (paracetamol 1gm/8 hours) till no fever and temperature less than 380c, and prophylactic anticoagulant low molecular weight heparin (enoxaparin 40/24 hours), prophylactic stress ulcer (pantoprazole 40mg/24hours)
  Other Names: Standard sepsis treatment

SUMMARY:
Sepsis is a leading cause of morbidity and mortality in intensive care units. Sepsis is a life-threatening organ dysfunction linked to a dysregulated host response to infection. It leads to overwhelming of systemic inflammation causing release of proinflammatory cytokines, which trigger overproduction of reactive oxygen species. Several animal studies with sepsis proved the effectiveness of montelukast and coenzyme Q10 as anti-inflammatory and antioxidants in preventing end organ damage, deterioration, and reducing mortality. Therefore, a clinical trial will be carried out to compare the efficacy and safety of montelukast versus co enzyme Q10 on the clinical outcome in patients with sepsis.

DETAILED DESCRIPTION:
Sepsis is now defined as a life-threatening organ dysfunction linked to a dysregulated host response to infection. This organ dysfunction can be identified using the Sequential Organ Failure Assessment (SOFA). Sepsis is a leading cause of morbidity and mortality in the intensive care unit (ICU). It has been reported that the short-term mortality rate ranges from 30 to 50%, depending on illness severity. The global epidemiological burden of sepsis is, however, difficult to ascertain. It is estimated more than 30 million people are affected by sepsis every year worldwide, resulting in potentially 6 million deaths annually. The mortality rate estimated to be 30% in sepsis and 80% in septic shock in the USA, and 12.8% in sepsis and 45.7% in septic shock in Europe. Reduced rates of reporting may influence estimations in developing countries.

Sepsis is characterized by overwhelming systemic inflammation causing a release of proinflammatory cytokines. The presence of infection leads to initial activation of the innate immune response. The resulting pro-inflammatory host response is both complex and redundant, involving many soluble inflammatory mediators, including cytokines [e.g., tumor necrosis factor (TNF) α and interleukin (IL) 6] and reactive oxygen/nitrogen species (e.g., nitric oxide (NO) and peroxynitrite), as well as multiple cell types, including neutrophils, macrophages, platelets, and endothelial cells. The up regulation of pro- and anti-inflammatory pathways leads to a system-wide release of cytokines, mediators, and pathogen-related molecules, resulting in activation of coagulation, and complement cascades, the resulting inflammation leads to progressive tissue damage, finally causing multi-organ dysfunction.

Sepsis-induced mitochondrial damage or dysfunction can result in cellular metabolic disorders, insufficient energy production, and oxidative stress, which give rise to the apoptosis of organ cells and immune cells, thus ultimately generate immune disorders, multiple organ failure, and even death. As during sepsis limited amount of oxygen supply, the free radical production increases dramatically while the machinery of the antioxidant system becomes damaged. Activated leukocytes release inflammatory cytokines, which trigger overproduction of reactive nitrogen species (RNS) and nitrogen oxide. Nitrogen oxide can bind to reactive oxygen species (ROS) peroxides to form RNS, which unfortunately brings about further damage to mitochondria, including mitochondrial, and mitochondrial DNA damage.

Hence, different treatment strategies have focused in minimizing this inflammatory syndrome without reaching a consensus. Numerous anti-inflammatory and antioxidants therapies have been proposed and studied, including corticosteroids, anti-cytokine approaches, selenium, vitamin C, as well as other various basic research-driven therapies.

Montelukast is a cysteinyl leukotriene receptor antagonist with anti-inflammatory and antioxidant properties. Cysteinyl leukotrienes (CysLTs) are formed by inflammatory cells, such as mast cells, eosinophils, and basophils. CysLTs are potent pro-inflammatory mediators that increase microvascular permeability and are effective chemotactic agents. CysLT receptors are present in the airways, liver, and other organs. CysLT1 antagonists, such as Montelukast, have been reported to ameliorate experimental colitis, burn- and sepsis-induced multi-organ damage. Montelukast acts by inhibiting neutrophil infiltration, balancing oxidant-antioxidant status, and controlling inflammatory mediator generation. Montelukast possesses anti-inflammatory effect through the inhibition of TNF-alpha stimulated by IL-8 expression through changes in nuclear factor-Kb, and the antioxidant effect is due to decreasing the ROS, and reactive nitrogen species (e.g. NO) production, and hence it could help ameliorate inflammation associated with sepsis.

Several studies reported montelukast as a safe and tolerable medication. It was reported in 1996 that the administration of 10 mg orally, montelukast to healthy adult patients, was well tolerated. Four years later, Storms and colleagues published safety data from 11 multicenters, randomized, controlled montelukast phase, which included numerous adult and pediatric patients. They reported that the administration of montelukast over 5 months as 200 mg/day, which is 20 times higher than the recommended clinical dose, was also tolerable and similar to placebo.

Many experimental model studies showed how montelukast is effective against sepsis. Şener and his colleagues postulated that montelukast possesses an anti-inflammatory effect on sepsis-induced hepatic and intestinal damage and protects against oxidative injury by a neutrophil-dependent mechanism. Another study concluded that montelukast treatment after Cecal Ligation and Puncture-Induced Sepsis potentially reduced mortality in experimental sepsis that was attributed to the reduction of organs' oxidative stress and the decrease in plasma cytokine levels. It was found also that montelukast might have cardioprotective effects against the inflammatory process during endotoxemia. This effect was attributed to its antioxidant and/or anti-inflammatory properties.

Coenzyme Q10 (Co enzyme Q10) is a fat-soluble molecule, naturally found in the diet and synthesized endogenously by all cells of our body in the mitochondrial inner membrane, that exists both in oxidized form (ubiquinone) and reduced form (ubiquinol). Co enzyme Q10 plays an essential role in the electron transport chain of mitochondria as the carrier of electrons from complex I and II to complex III. Disruption of this mechanism can compromise oxidative phosphorylation, thereby leading to decreased levels of cellular energy (adenosine triphosphate (ATP)) production. Previous studies have reported that Co enzyme Q10 (Co enzyme Q10) can prevent the start and diffusion of lipid peroxidation, scavenge free radicals, and decrease pro-inflammatory cytokine production. The deficiency of Co enzyme Q10 induced by mitochondrial failure in sepsis may play a role in hypoxia, oxidative organ damage, hypo-perfusion, and ultimately leading to death. There is considerable evidence from randomized controlled clinical studies that Co enzyme Q10 can ameliorate such inflammation, via effects on circulatory pro-inflammatory markers such as C-reactive protein (CRP), interleukins 1 and 8 (IL-1, IL-8), and tumor necrosis factor-alpha (TNF).

CoenzymeQ10 showed its activity against sepsis in many previous studies. Coenzyme Q10 administered during the hypodynamic phase of sepsis decreased splenic, renal and cardiac damage and organ damage. It also assisted in the reduction of septic liver injury as indicated by the upregulation of beclin 1 as well as the suppression of AST, ALT, ALP, p62, IL-6, TNF-α, NLRP 3, and IL-1β as reported in another animal study. Moreover, it has been reported that critically ill patients had lower levels of CoenzymeQ10 levels on ICU admission compared to healthy controls and exhibited a further decrease in sepsis and septic shock. Donnino and colleagues provided original data suggesting a CoenzymeQ10 deficiency in patients with septic shock, and this is a new step toward a study testing CoenzymeQ10 as a potential therapeutic agent for patients with septic shock

ELIGIBILITY:
Inclusion Criteria:

Age >18 years old.

* Males and females
* Confirmed diagnosis of sepsis according to the third sepsis definition which include documented or suspected infection, plus an acute change in total SOFA score ≥ 2 points

Exclusion Criteria:

* Pregnancy
* A severe moribund state
* An anticipated ICU stay of less than 24 hours.
* Patients with a history of hypersensitivity to montelukast or co enzyme Q10.
* Patients with systemic eosinophilia in the blood or vasculitis.
* Patients with neuropsychiatric diseases as hallucinations, depression or suicidal thoughts that put the patient at risk when participating in the study.
* Unable to receive enteral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Twenty-eight-day mortality | Starting from the randomization date up to 28 days
  All patients will be followed up in the ICU and by phone calls after discharge. The 28-day mortality rate will be evaluated and recorded.

SECONDARY OUTCOMES:
Sequential organ failure assessment score | Starting from the randomization date,on day 3, on day7, and then every 3 days till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  It measures sepsis related end organ damage. It includes serum creatinine level as the renal component, total bilirubin level as the hepatic component, Glasgow coma score as the central nervous system component, mean arterial pressure, PaO2, and platelet count.
  The minimum value is zero, and the maximum value is 24, the higher the score, the worse the outcome, as the maximum value means the expected mortality is more than 90%, and the minimum value means the expected mortality is less than 10%
C- reactive protein | Starting from the randomization date,on day 3, and on day7
  Marker C- reactive protein will evaluate the state of inflammation in septic patients.
Heart rate | Starting from the randomization date till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  Heart rate will be monitored and recorded for septic patients
ICU length of stay | Starting from the randomization date till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  Length of patient stay in the ICU.
Length of hospital stay | Starting from the randomization date till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  Length of patient stay in the hospital.
The need for mechanical ventilation The number of patients who will need mechanical ventilation in addition to the duration of ventilation will be recorded | Starting from the randomization date till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  The number of patients who will need mechanical ventilation in addition to the duration of ventilation will be recorded
The need for vasopressors | Starting from the randomization date till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  The number of patients who will receive vasopressors in addition to the dose and duration of vasopressor use will be recorded.
The incidence of treatment side effects and the number of their occurrence | Starting from the randomization date till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  Record the incidence of treatment side effects and the number of their occurrence including dermatological reactions, nausea, vomiting or diarrhea, cough or acute bronchitis, headache, gastrointestinal disorders, fatigue, gastrointestinal upset, and heartburn.
Serum tumor necrosis factor α level | Starting from the randomization date, and on day 7
  An inflammatory marker
Serum MDA level | Starting from the randomization date, and on day 7
  An oxidative stress marker
Temperature | Starting from the randomization date till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  Temperature will be recorded for septic patients
Blood pressure | Starting from the randomization date till patient ICU discharge or death from any cause, which comes first, assessed up to 30 days.
  Both systolic and diastolic blood pressures will be monitored and recorded for septic patients

CONTACTS AND LOCATIONS:
Overall Officials: Salwa om Amin, PHD, Principal Investigator — Ain Shams University
Locations (1):
- Ghada El Adly, Cairo, Egypt

REFERENCES:
- [Derived] Eladly GH, Amin SOE, Sabri NA, Shawki MA. The clinical outcome of Montelukast versus co-enzyme Q10 in adult patients with sepsis: A randomized controlled clinical trial. J Crit Care. 2026 Feb;91:155225. doi: 10.1016/j.jcrc.2025.155225. Epub 2025 Aug 21. PMID 40845766